CLINICAL TRIAL: NCT04227665
Title: Identification of Biological Markers for Hypoxic Exposure and Use of Recombinant Human Erythropoietin
Brief Title: Identifying Biological Markers for Altitude Exposure and Use of Recombinant Human Erythropoietin (rHuEPO)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: World Anti-Doping Agency (Other); German Sport University, Cologne (Other); Universidad de Granada (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Nikolai Nordsborg, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: H-17036662
Record Dates: First submitted 2018-05-07; First posted 2020-01-14 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — Sea Level Rise; Altitude

STUDY DESIGN:
Intervention Model Description: Explorative design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sea level (Experimental): Sea level training camp
  Interventions: Other: Sea level
- Altitude (Experimental): Altitude training camp
  Interventions: Other: Altitude

INTERVENTIONS:
Other: Sea level — Sea level exposure / sea level exposure combined with microdoses of rHuEPO
  Arms: Sea level
Other: Altitude — Altitude exposure / altitude exposure Iron metabolism
  Arms: Altitude

SUMMARY:
The project represents a well powered study of the human response to altitude exposure combined with rHuEPO treatment. A total of 20 male and 20 female non-competing athletes will participate. The participants will be exposed to a period of hypobaric hypoxia at 2.320 m for four weeks and a sea-level intervention period of four weeks. The participants will be blinded and randomly allocated to intra venous injection with 20 IU per kg body weight of recombinant human erythropoietin or placebo every second day for the initial three weeks of each intervention. Included subjects will be runners due to the good possibility of recruitment and conduction of training at altitude. Samples are collected weekly for four weeks prior to each intervention period, during the four week intervention and four weeks after. This approach yields a highly valuable biobank for identification of markers sensitive to initiation of rHuEPO injections as well as termination of injections.

DETAILED DESCRIPTION:
The main hypothesis for this study is that metabolomics and proteomics methods can identify biomarkers that are sensitive to altitude exposure and recombinant human erythropoietin treatment, respectively. Secondarily, the hypothesis is that the identified biomarkers can distinguish between altitude exposure and abuse of rHuEPO.

We will include 20 Danish men and 20 Danish women aged 18-35 years. The inclusion criteria are a maximum oxygen uptake rate (VO2max) > 48 ml / kg / min for men and > 43 ml / kg / min for women. All trial participants must have > 2 years of history in regular exercise including running (> 2 times a week; > 30 min per session) and capable of performing a 5 km run in 22 min for men and 25 min for women at sea level on a level surface in dry conditions and a temperature between 10 and 20 degrees C. Furthermore, the participants must not have experienced running related injuries within the past two years.

The experimental protocol consists of two experimental periods, both of which must be performed by all participants. Both periods contain a baseline period of four weeks followed by four weeks training camp and four weeks follow up. The training camp in one period of experiments is performed at sea level while the training camp in the other period is performed at 2320 m above sea level. Each period is separated by a minimum of two months to ensure that the participants have returned to baseline values. During the two intervention periods, the participants will be transported by air and car to the destination of the respective training camp. It is expected that the participants train for 1-2 hours a day on average and that the time spent for the measurements described is ~ 5-7 hours a week.

To investigate whether the described methods can identify sensitive biomarkers for the physiological response due to rHuEPO treatment, the participants will be treated with rHuEPO.

The distribution of participants allows the following:

* 28 participants receive rHuEPO at sea level, thereby identifying biomarkers sensitive for use of rHuEPO
* 28 participants receive placebo under altitude exposure, whereby biomarkers sensitive to altitude exposure can be identified
* 12 participants receive placebo at sea level, whereby random fluctuations of the identified biomarkers can be determined.
* 12 participants receive rHuEPO under altitude exposure, whereby the identified rhuEPO biomarkers and altitude exposure can be tested for whether they can be used to separate individuals receiving rHuEPO under altitude exposure from individuals receiving placebo under altitude exposure.
* 8 participants receive placebo at sea level and altitude exposure, whereby natural and random individual fluctuations can be determined over a longer period (> 6 months). Since random individual fluctuations can be determined at n = 1, n = 8 will be sufficient to determine this.

ELIGIBILITY:
Inclusion Criteria:

* Male: VO2max > 48 ml/min/kg bodyweight and 5km run < 22 min, Female: VO2max > 43ml/min/kg bodyweight and 5km run < 25 min A minimum of 2 years injury running training

Exclusion Criteria:

* Age, insufficient fitness or injury

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Identification of metabolites in urine for rHuEPO and altitude exposure | 5 years
  Urine is analyzed by metabolomics and the metabolites for rHuEPO and altitude are verified using an exploratory design.
  More specifically, the aim is to identify the resulting metabolites from altitude exposure and treatment with rHuEPO as these are not yet known In this WADA-supported research project, the aim is to identify high sensitivity biomarkers for altitude exposure through a metabolomics methods, as 'omics' methods have previously shown promising results in other exposure contexts. However, being the first of its kind in antidoping the resulting metabolites from rHuEPO misuse and altitude have not yet been identified. Thus, an exact description of these is not possible
Identification of human metabolites in serum for rHuEPO and altitude exposure | 5 years
  Human serum is analyzed by metabolomics and the metabolites for rHuEPO and altitude are verified using an exploratory design.

SECONDARY OUTCOMES:
Reticulocyte percentage | Up to 24 weeks
  Reticulocyte percentage, will be measured to determine variation as a result of either 12 weeks exposure to altitude or sea-level (24 weeks in total).
Hemoglobin concentration | Up to 24 weeks
  [hemoglobin] will be measured to determine variation as a result of either 12 weeks exposure to altitude or sea-level.
OFF-score | Up to 24 weeks
  OFF-score (computed from reticulocyte perscentage and hemoglobin concentration), will be measured to determine variation as a result of either 12 weeks exposure to altitude or sea-level.
Maximal oxygen uptake (VO2max) | Up to 24 weeks
  VO2max (ml/min) measured by incremental work load on a treadmill
Iron metabolism | Up to 24 weeks
  Markers of iron metabolism such as hepcidin and erythroferrone are collected analyzed for evaluation of iron metabolism during and after a training camp at 2300m above sea level
Work economy | Up to 24 weeks
  Running efficiency (%) measured by energy expenditure on a treadmill
Sustainable workload | Up to 24 weeks
  Lactate threshold (mmol/L) measured on a treadmill
Running performance | Up to 24 weeks
  5000m time trial performance (time) measured on a 400m running track
Muscle oxygenation | Up to 24 weeks
  Muscle oxygenation measured by near-infrared spectroscopy during running on a treadmill
Total hemoglobin mass | Up to 24 weeks
  Total hemoglobin mass will be measured by two-minute carbon-monoxide re-breathing to determine variation as a result of either 12 weeks exposure to altitude or sea-level.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bejder, Msc, Principal Investigator — Universuty of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Copenhagen Ø, Denmark

IPD SHARING:
Plan to Share IPD: No
Fully anonymous data will be shared with other researchers.

REFERENCES:
- [Derived] Arrebola-Moreno AL, Casuso RA, Bejder J, Bonne TC, Breenfeldt Andersen A, Aragon-Vela J, Nordsborg NB, Huertas JR. Does Hypoxia and Stress Erythropoiesis Compromise Cardiac Function in Healthy Adults? A Randomized Trial. Sports Med Open. 2022 Nov 5;8(1):137. doi: 10.1186/s40798-022-00531-x. PMID 36334130